CLINICAL TRIAL: NCT02504684
Title: Endovenous Laser Ablation of the Great Saphenous Vein Comparing 1920-nm and 1470-nm Diode Laser
Brief Title: Treatment of Saphenous Vein Reflux With 1920-nm Diode Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Vascular BH (Other)
Responsible Party: Principal Investigator, Daniel Mendes Pinto, Daniel Mendes Pinto, MD, Instituto Vascular BH
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20130220
Record Dates: First submitted 2015-07-15; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Varicose Veins
Keywords: varicose veins; endovenous laser treatment; endovenous thermal ablation; saphenous vein
MeSH Terms: conditions — Varicose Veins | interventions — Lasers, Semiconductor; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1470-nm (Active Comparator): Endovenous 1470-nm diode laser
  Interventions: Device: Endovenous 1470-nm diode laser
- 1920-nm Group (Experimental): Endovenous 1920-nm diode laser
  Interventions: Device: Endovenous 1920-nm diode laser

INTERVENTIONS:
Device: Endovenous 1920-nm diode laser — Patients with saphenous veins treated with a new 1920-nm diode endolaser.
  Other Names: 1920-nm laser
  Arms: 1920-nm Group
Device: Endovenous 1470-nm diode laser — Patients with saphenous veins treated with the standard 1470-nm diode endolaser.
  Other Names: 1470-nm laser
  Arms: 1470-nm

SUMMARY:
Objective: Compare venous occlusion rates at a one-year follow-up comparing 1920-nm versus 1470-nm laser treatment. Design: Non-randomized prospective study. Methods: Adult patients with varicose veins associated with great saphenous reflux were included. Procedures were performed between February and April of 2013. The 1470-nm laser ablation was performed in continuous mode, power being set between 8 and 10 W, while for the 1920-nm it was set between 5 and 6 W. Checking for vein closure was performed during the thermal ablation procedure, LEED (linear endovenous energy density) being calculated after the procedure. Follow-up data were collected at the 7-day, 30-day, 3-month, 6-month and 1-year visits, and involved clinical and ultrasound evaluation, measurement of occlusion extent.

DETAILED DESCRIPTION:
INTRODUCTION The treatment of varicose veins secondary to saphenous vein reflux has undergone a major shift in the past decade, primarily led by the introduction of less invasive techniques. Wavelengths of 810, 940 and 980 nm have higher rates of absorption by hemoglobin. Water chromophore is associated with an initial energy absorption peak at 980 nm, followed by peaks at 1500 and 2000 nm. The energy released into the vein lumen is therefore absorbed by water as well as by cellular and interstitial proteins. In contrast, laser beams with longer wavelengths act more specifically on water absorbance, resulting in less energy expenditure, such as in the case of the 1470-nm diode endolaser. An endoluminal energy density (LEED) around 50-160 J/cm has been demonstrated to effectively lead to venous occlusion, although LEEDs above 100 J/cm can also be associated with higher complication rates. In contrast, the 1920-nm diode laser is more specific for water and hemoglobin chromophores, tissue absorption at this wavelength being at least 2.5 times greater than the one obtained with the 1470-nm laser. It is therefore expected that less energy would be required to generate the same amount of venous closure.

The aim of this study is to compare diode 1920-nm versus 1470-nm laser in the treatment of great saphenous vein reflux. The primary outcome was venous segment occlusion at the one-year follow-up. Secondary outcomes included LEED, postoperative complications, and clinical outcomes measured through the Clinical, Etiology, Anatomical and Pathological classification (CEAP), the Venous Clinical Severity Score (VCSS) and a patient satisfaction scale.

METHODS This is a prospective study to evaluate the results of the 1920-nm vs. 1470-nm laser. Patients agreeing to participate were offered informed consent, recruitment occurring between February and April of 2013. Participants enrolled between February and mid-March of 2013 underwent treatment with the 1470-nm laser, while those enrolled between mid-March and April underwent treatment with the 1920-nm laser.

Patients between 18 and 70 years old who had varicose veins associated with reflux of the great saphenous veins were included. The exclusion criteria were: patients with a previous history of thrombophlebitis, deep vein thrombosis or who had undergone any previous surgery for this condition, thermal ablation or sclerotherapy. For bilateral cases, both limbs were treated during the same surgical session.

Data on clinical history, physical examination, CEAP classification, VCSS (Venous Clinical Severity Score) and VDS (Venous Disability Score) were collected. The extent of the great saphenous reflux was measured along with its main diameter at the level of the saphenofemoral junction as well as at the knee level. Reflux was defined as retrograde when reaching a speed greater than 3 cm/second during a Valsalva maneuver or through leg compression maneuvers.

All patients underwent procedures under spinal anesthesia. The great saphenous vein was punctured at the most distal point of reflux and a 6F introducer was positioned. All cases were conducted with a 600-micron radial fiber positioned between 2.0 and 3.0 cm from the saphenofemoral junction. A tumescence with 0.9% saline solution was placed under ultrasound guidance around the full length of the saphenous vein. All patients were in a 30-degree Trendelenburg position. Surgical procedures involved the saphenous ablation and phlebectomy.

Saphenous ablation with a 1470-nm laser was performed in continuous mode, with a power of 8 to 10 W, determined as a function of the diameter of the vessel as well as surgeon's preference. The 1920-nm laser was also used in continuous mode, with 5 to 6 W power. Vein closure monitoring during the thermal ablation procedure was conducted through ultrasound while pulling-off the fiber. At the end of the procedure, the total amount of energy used in each limb was recorded for LEED calculation, measured as total energy used in the limb (J) over vein length (cm).

First follow-up occurred at postoperative week one, with subsequent evaluation at 30 days, three months, six months and one year. At each assessment, symptoms were recorded and an ultrasound evaluation was performed. Patient satisfaction was evaluated at 1-week through the following questions "Are you satisfied with your surgery?" and "Would you choose the same treatment again?" Both questions were presented as a Likert scale where 0 = very satisfied, 1 = satisfied, 2 = indifferent, 3 = not satisfied, 4 = very dissatisfied.

The primary endpoint for this study was the percentage of occluded venous segments at the 6-month follow-up. Extension of the occluded saphenous vein segment was measured at each visit through a tape guided by ultrasound to determine occlusion points. A segment was considered patent if it was compressible and with reflux after muscle compression in a standing position. The length of the occluded vein segment was compared with the length of the segment where thermal ablation was performed, thus allowing us to calculate the segment closure percentage. Secondary end-points were the presence of ecchymosis, induration, paresthesia, skin burns and deep vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with varicose veins associated with reflux of great or small saphenous veins

Exclusion Criteria:

* Patients under 18 years old or over 70 years.
* Acute or previous thrombophlebitis or deep vein thrombosis.
* Pregnant patient.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Venous segment occlusion at one-year follow-up | one year
  Extent of venous occlusion measured in centimeters. The length of occluded vein segment is measured and compared with total extension of the vein treated with the endolaser.

SECONDARY OUTCOMES:
Ecchymosis extension | 7 days
  Extent of ecchymosis noticed after endolaser treatment of the saphenous veins measured in centimeters and compared to the total extension of vein treated with the endolaser.
Presence of induration | 30 days
  Induration noticed on the saphenous vein path.
Presence of Paresthesia | 30 days
  Presence or absence of paresthesia in the limb treated by endovenous laser
Skin burns | 7 days
  Presence or absence of skin burns in the limb treated by a endovenous laser
Deep vein thrombosis | 7 days
  Presence or absence of deep vein thrombosis diagnosed by ultrasound in the limb treated by endovenous laser

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Pinto, MD, Principal Investigator — Instituto Vascular BH
Locations (1):
- Children ABC hospital, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Result] Rasmussen LH, Lawaetz M, Bjoern L, Vennits B, Blemings A, Eklof B. Randomized clinical trial comparing endovenous laser ablation, radiofrequency ablation, foam sclerotherapy and surgical stripping for great saphenous varicose veins. Br J Surg. 2011 Aug;98(8):1079-87. doi: 10.1002/bjs.7555. PMID 21725957
- [Result] Siribumrungwong B, Noorit P, Wilasrusmee C, Attia J, Thakkinstian A. A systematic review and meta-analysis of randomised controlled trials comparing endovenous ablation and surgical intervention in patients with varicose vein. Eur J Vasc Endovasc Surg. 2012 Aug;44(2):214-23. doi: 10.1016/j.ejvs.2012.05.017. Epub 2012 Jun 15. PMID 22705163
- [Result] Pan Y, Zhao J, Mei J, Shao M, Zhang J. Comparison of endovenous laser ablation and high ligation and stripping for varicose vein treatment: a meta-analysis. Phlebology. 2014 Mar;29(2):109-19. doi: 10.1177/0268355512473911. Epub 2013 May 6. PMID 23390218
- [Result] Vuylsteke ME, Vandekerckhove PJ, De Bo T, Moons P, Mordon S. Use of a new endovenous laser device: results of the 1,500 nm laser. Ann Vasc Surg. 2010 Feb;24(2):205-11. doi: 10.1016/j.avsg.2009.06.024. Epub 2009 Sep 11. PMID 19748212
- [Result] von Hodenberg E, Zerweck C, Knittel M, Zeller T, Schwarz T. Endovenous laser ablation of varicose veins with the 1470 nm diode laser using a radial fiber - 1-year follow-up. Phlebology. 2015 Mar;30(2):86-90. doi: 10.1177/0268355513512825. Epub 2013 Nov 29. PMID 24291781